CLINICAL TRIAL: NCT05994118
Title: Exploring the Role of Physiological, Cognitive, and Personal Features in the Link Between Placebo-effect and Variability of Pain Reports
Brief Title: Physiological, Cognitive, and Personal Features in the Link Between Placebo-effect and Variability of Pain Reports
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Haifa (Other)
Collaborators: Western Galilee Hospital-Nahariya (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 0044-20-NHR
Record Dates: First submitted 2022-04-13; First posted 2023-08-16 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Chronic Back Pain
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: Subcutaneous injection of Saline solution (NACL 0.9%) in the buttock
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal Saline (Placebo Comparator): 0.5 milliliter of NACL 0.9% subcutaneous saline injection
  Interventions: Other: NaCl 0.9% (normal saline)
- Magnetized Normal Saline (Active Comparator): 0.5 milliliter of magnetized NACL 0.9% subcutaneous saline injection
  Interventions: Other: Magnetized Normal Saline

INTERVENTIONS:
Other: NaCl 0.9% (normal saline) — Subcutaneous normal saline injection
  Arms: Normal Saline
Other: Magnetized Normal Saline — Magnetized Normal Saline
  Arms: Magnetized Normal Saline

SUMMARY:
This study attempt to identify whether and how factors known or considered to be related with analgesic placebo effect or variability of pain reports separately, may contribute to their coupling. Among these factors - personal traits such as optimism, focus of attention, suggestibility, and short-term memory along with characteristics of stress and relaxation. Additionally, the role of pain sensitivity and the individual's pain modulation profile in the relationship between analgesic placebo effect and variability of pain reports will be examined.

DETAILED DESCRIPTION:
Data will be collected from 130 patients with non-specific chronic back pain that will be recruited for a prospective cross-sectional study. To characterize the main study variables, the participants will undergo the Focused analgesia selection test (FAST) which evaluates within-subjects variability of pain reports, and placebo manipulation containing administration of an inert injection accompanied by a verbal suggestion, which is expected to produce placebo effects. The involvement of additional factors considered associated with the within-subjects variability of pain reports and the placebo response will be explored. Stress and well-being characteristics will be examined by measuring cortisol levels in saliva and in hair, salivary level of Secretory Immune globulin A (SIgA), and an autonomic nervous system function and a stress perception questionnaire. Personal traits such as suggestibility, optimism, and Focus of attention, will be examined using questionnaires. Memory will be assessed by memory task, and factors related to the pain modulation system will be examined using psychophysical tests, and a pain sensitivity questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Literate adults
* Aged 18 - 80 years
* A diagnosis of chronic back pain
* Sufferings from back pain during the last 3 months or more, with an intensity of 3 or more on a 0-10 NRS

Exclusion Criteria:

* Mental retardation or cognitive impairment
* Pregnancy or breast-feeding
* Malignancy and a diagnosis of malignant disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-03-21 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Reduction of pain following placebo injection | Half an hour after injection
  The reduction in pain intensity on the 0-100 numerical rating scale (NRS) after normal saline injection
Within-subjects variability of day-to-day clinical pain reports | 7 days before study visit
  The variance of within person pain scores reported on a 0-100 Visual Analog Scale VAS during 7 days via pain-dairy at baseline

SECONDARY OUTCOMES:
The Focused Analgesia selection task (FAST) | Once, at baseline
  Experimental paradigm which allow calculation of within-subjects variability of pain reports in response to thermal stimuli

OTHER OUTCOMES:
Pain modulation - Temporal Summation | Once, at baseline
  Change in pain intensity on the 0-100 numerical rating scale (NRS) in response to the first and last electrical noxious stimuli
Pain modulation - Conditioned pain modulation | Once, at baseline
  Change in pain intensity on the 0-100 numerical rating scale (NRS) in response to concurrent noxious stimuli
Biological markers - cortisol | 1 day (Before and after administration of saline)
  Saliva cortisol levels
Biological markers - secretory IgA | 1 day (Before and after administration of saline)
  Saliva secretory IgA level
Biological markers - oxytocin | 1 day (Before and after administration of saline)
  Saliva oxytocin level
Autonomic measures - Heart rate variability | 1 day (Before and after administration of saline)
  As measured by a monitor
Autonomic measures - blood pressure | 1 day (Before and after administration of saline)
  As measured by a monitor
Short-term memory | Once, at baseline
  via the Digit Span test
Pain sensitivity via QST | 1 day (Before and after administration of saline)
  Mechanical pain thresholds
Questionnaire - Optimism | Once, at baseline
  Via the life orientation test revised (LOT-R)
Questionnaire - pain sensitivity | Once, at baseline
  Via the pain sensitivity questionnaire (PSQ)
Questionnaire - interoceptive awareness | Once, at baseline
  Via the Multidimensional assessment of interoceptive awareness (MAIA questionnaire)
Questionnaire - direction of attention | Once, at baseline
  Via the Self consciousness scale revised
Questionnaire Body awareness | Once, at baseline
  via the body awareness Questionnaire (BAQ)
Questionnaire - suggestibility | Once, at baseline
  Via the short suggestibility scale (SSS)
Questionnaire - expectations | Once, at baseline
  via the expect Questionnaire
Questionnaire - perceived stress | Once, at baseline
  via the perceived stress scale

CONTACTS AND LOCATIONS:
Overall Officials: Roi Treister, PhD, Principal Investigator — University of Haifa
Locations (1):
- Galilee Medical center, Nahariya, Israel

IPD SHARING:
Plan to Share IPD: Yes
Once published, the data (without any personal identification) will be available upon request